CLINICAL TRIAL: NCT03635372
Title: A Comparison of Effectiveness of Oral Sucrolfate, Alginate and Hydrotalcide in Dispeptic Pain Treatment: Randomized Trial
Brief Title: A Comparison of Effectiveness of Oral Sucrolfate, Alginate and Hydrotalcide in Dispeptic Pain Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Bulent Erdur, professor, Pamukkale University
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 2016TPF001
Record Dates: First submitted 2018-08-15; First posted 2018-08-17 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Dyspepsia
Keywords: Dyspepsia; Emergency Department; Antacid; Viscous Lidocaine
MeSH Terms: conditions — Dyspepsia; Emergencies | interventions — Alginates; Sucralfate; hydrotalcite

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Alginate (Experimental): 10 cc of Alginate peroral
  Interventions: Drug: Alginate
- Sucralfate (Experimental): 10 cc of Sucralfate peroral
  Interventions: Drug: Sucralfate
- Hydrotalcite (Experimental): 10 cc of Hydrotalcite peroral
  Interventions: Drug: Hydrotalcite

INTERVENTIONS:
Drug: Alginate — 10 cc of Alginate peroral
  Other Names: Gaviscon Lipuid
  Arms: Alginate
Drug: Sucralfate — 10 cc of Sucralfate peroral
  Other Names: Antepsin Suspension
  Arms: Sucralfate
Drug: Hydrotalcite — 10 cc of Hydrotalcite peroral
  Other Names: Talcid Suspension
  Arms: Hydrotalcite

SUMMARY:
Dyspepsia is a very common but non-specific complaint that may indicate a group of symptoms that can be attributed to the upper gastrointestinal system, such as epigastric discomfort, abdominal bloating or fullness, stomach upset and nausea or vomiting that may be associated with food.

This study aimed to improve treatment management of patients with complaints of dyspeptic pain and emergency services, and to compare treatment efficacy of oral sucralfate, alginate and hydrotalcite, which are widely used in our country. Literature According to our research, our study is the first study to compare different antacids in our study of emergency serviste dyspepsia.

DETAILED DESCRIPTION:
This study was performed prospectively, randomly, controlled, double-blind to compare the efficacy of oral sucralfate, alginate and hydrotalcite in patients presenting with emergency department dyspeptic complaints at Pamukkale University Medical Faculty Hospital Emergency Medicine Department.

Patients who were referred to the emergency department with stomach ache or dyspeptic complaints were taken to the study. Treatment medicines were applied according to the randomization scheme of the study patients.

This study was carried out in Pamukkale University Faculty of Medicine Emergency Medicine Department during 8 months between 01.03.2016 and 30.10.2016. Approximately 98,000 adult patients / year in the emergency department have a research assistant and / or faculty member who will check the research as a 24-hour primer. This study included 300 cases between 18 and 60 years of age who were admitted to our emergency department with dispeptic complaints, agreed to participate in the study, informed consent, and met inclusion criteria. The criteria for receiving and not receiving work were specified at the beginning of the study.

When appropriate patients were admitted to the study, the patient was taken to the emergency monitoring monitor and monitored once the written consent was obtained. Patients were assigned to one of the study groups according to the study number, according to the randomization scheme prepared by a non-emergency service computer. The numbers for the previously numbered workgroups were kept in unmarked envelopes and the envelope was opened by the study nurse to prepare the study medicine. The study medicines were prepared by an independent person who did not participate in the study or by the responsible work nurse who was at the helpline and was given to the patient by the other nurse. For each group, the drugs prepared in a 10 cc syringe were wrapped around the syringe with a color patch that did not show any similarity. When the medication was given to the patient, the patient's nose was closed and the drug smell was not taken. Patients were observed for 30 minutes in the emergency department and 30-minute VAS (Visual Analog Scale) score 5 and above were given to the patient for rescue treatment.

The information and data of the patients were collected by questionnaire. In the first part of the questionnaire, patients' demographic information address, telephone numbers, medical backgrounds, medications and vital findings were recorded. Detailed physical examinations of all patients were evaluated by emergency physician. Patients diagnosed with dyspepsia other than dyspepsia such as acute coronary syndrome, pancreatitis, cholecystitis, acute abdomen, ileus, malignancy and gastroenteritis were excluded as a result of history and physical examination. Patients who did not give their consent to participate were also excluded from the study. The patient with unexplained dyspepsia was directed to the gastroenterology polyclinic for endoscopy with necessary information. After discharge, patients were asked whether they had recurring epigastric pain within 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* Stomach pain, swelling or dispeptic complaints.
* Men and women between the ages of 18-60.
* Patients with VAS> 5.

Exclusion Criteria:

* Pregnancy and lactation.
* Sucralfate, alginate, hydrotalcite allergy.
* Emergency service arrives with acute psychiatric symptoms.
* Gastrointestinal system bleedings.
* Chronic renal failure, liver cirrhosis, structural and functional heart disease.
* Gastric malignancy and terminal illness.
* Patients suspected of having a different problem such as ileus, biliary colic,
* pancreatitis, hepatitis.
* Patients who refuse to participate in the study.
* Those who can not use VAS.
* Presence of ischemic findings on the arrival ECG.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2017-06-20 (Actual); Primary Completion 2017-10-22 (Actual); Study Completion 2017-11-25 (Actual)

PRIMARY OUTCOMES:
Relief of Gastric Pain | Change from baseline in dispeptic complaint VAS scores at 60 minutes
  Compare relief of dispeptic complaint with using VAS (Visual Analog Scale) in 3 groups of alginate, sucralfate and hydrotalcite patients. Patients' pain scores were recorded using 0-100 mm VAS (Visual Analog Scale) to score the degree of dyspeptic complaints. VAS; It is composed of a measured horizontal or vertical line and often carries definitions of "no symptoms" on one end and "severe symptoms" on the other end. The patient is told to mark a point on the line according to the severity of the symptom. The location of the marker allows the severity of the symptom to be measured. The VAS markings on the evaluation forms prepared for the study before and during the procedure were made by the patient himself and regardless of the previous sign. Patients with VAS> 50 were treated. Patients were observed for 60 minutes in the emergency department and 60-minute VAS (Visual Analog Scale) score above 50 were given to the patient for rescue treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Gulgun Battal, MD, Principal Investigator — Pamukkale University
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No